CLINICAL TRIAL: NCT04342806
Title: Healthcare Worker Exposure Response and Outcomes (HERO) Registry Study
Brief Title: Healthcare Worker Exposure Response and Outcomes (HERO) Registry Study, COVID-19
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00105284
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Health Care Worker (HCW); COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HCWs currently working in the US, and their families and communities: The HERO Registry will include HCWs currently working across the United States, and their families and communities. For the purposes of this study, a "healthcare worker" is defined as an individual who currently works in a setting where individuals receive healthcare. (Note: individuals do not have to work directly with patients, but may have any role within a setting where individuals receive healthcare, such as housekeeping, food service, etc.)

SUMMARY:
The HERO Registry provides a resource for collecting information on Healthcare Workers (HCWs) currently working in the United States, and their families and communities. The overall goal of the Registry is to develop the infrastructure necessary to create and engage a community of people who may be eligible for participation in future research studies, including those of COVID-19 prophylaxis and treatment.

DETAILED DESCRIPTION:
The HERO Registry provides a resource for collecting information on Healthcare Workers (HCWs) currently working in the United States, and their family members and communities. The overall goal of the Registry is to create and engage a community of HCWs and their families and communities who may be eligible for participation in future research studies, including those of COVID-19 prophylaxis and treatment. The HERO registry will create a repository of adults interested in COVID-19 research that can be eligible for future research studies. The main objectives of the study are 1) create a virtual community of adult HCWs in the United States, and their families and communities, 2) Identify adults interested in engaging in upcoming research studies, including those related to COVID-19, and 3) Create a dataset of health related measurements, risk factors, and outcomes for future analysis. The population of interest is adult healthcare workers in the United States, and their families and communities.

All analysis of the HERO Registry will be exploratory in nature. Analysis may include descriptive statistics of the cohort, statistical associations between variables of interest, and predictive modeling for health outcomes and behaviors. Analyses may be conducted on all participants in the HERO Registry or may be conducted on subpopulations defined based on clinical, demographic or other factors.

There is no direct benefit to the participants for their participation in this study, but the information obtained will be used in scientific research and may be helpful to the participant or others in the future. Participants may experience indirect benefits such as learning about their own health, access to health data, and opportunities to participate in future research.

ELIGIBILITY:
Inclusion Criteria:

* A member of one of the following three groups:

  * Individual currently works in a setting where individuals receive healthcare ("healthcare worker") (including emergency medical services), OR
  * A family member of a healthcare worker, OR
  * A member of a healthcare worker's community
* Age ≥ 18
* Able to speak and read English or Spanish

Exclusion Criteria:

* There are no specific exclusion criteria for this study. Participants must meet inclusion criteria.

Ages: 18 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The HERO Registry will include HCWs currently working across the United States, and their families and communities. For the purposes of this study, a "healthcare worker" is defined as an individual who currently works in a setting where individuals receive healthcare. (Note: individuals do not have to work directly with patients, but may have any role within a setting where individuals receive healthcare, such as housekeeping, food service, etc.)
Sampling Method: Non-Probability Sample
Enrollment: 51466 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Number and percent of participants who enroll in the HERO Registry Study by geographic region, age, COVID-19 risk factors, and past COVID-19 diagnosis | Up to 79 years
Distribution of COVID-19 risk factors by participant characteristics | Up to 79 years
Proportion of participants undergoing changes in health status (e.g. new diagnosis of COVID-19, ER visits, hospitalization) | Up to 79 years
Proportion of all participants enrolled in the HERO Registry who participate in an ancillary research study | Up to 79 years
Proportion of participants who continue to supply information about their health to the HERO Registry at various time points after their enrollment | Up to 79 years

CONTACTS AND LOCATIONS:
Overall Officials: Emily O'Brien, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lusk JB, Manandhar P, Thomas LE, O'Brien EC. Association between characteristics of employing healthcare facilities and healthcare worker infection rates and psychosocial experiences during the COVID-19 pandemic. BMC Health Serv Res. 2024 May 24;24(1):659. doi: 10.1186/s12913-024-11109-6. PMID 38783301
- [Derived] Apple R, O'Brien EC, Daraiseh NM, Xu H, Rothman RL, Linzer M, Thomas L, Roumie C. Gender and intention to leave healthcare during the COVID-19 pandemic among U.S. healthcare workers: A cross sectional analysis of the HERO registry. PLoS One. 2023 Jun 16;18(6):e0287428. doi: 10.1371/journal.pone.0287428. eCollection 2023. PMID 37327216
- [Derived] Chen-Lim ML, McCabe MA, Xu H, Thomas LE, Forrest CB, Birnbaum S, Webb LE, O'Brien EC. Experiences of U.S. Nurses Compared With Nonnurses in the First Year of COVID-19: Findings From a National Registry. Nurs Res. 2022 Nov-Dec 01;71(6):421-431. doi: 10.1097/NNR.0000000000000610. Epub 2022 Jul 23. PMID 35878076
- [Derived] Forrest CB, Xu H, Thomas LE, Webb LE, Cohen LW, Carey TS, Chuang CH, Daraiseh NM, Kaushal R, McClay JC, Modave F, Nauman E, Todd JV, Wallia A, Bruno C, Hernandez AF, O'Brien EC; HERO Registry Research Group. Impact of the Early Phase of the COVID-19 Pandemic on US Healthcare Workers: Results from the HERO Registry. J Gen Intern Med. 2021 May;36(5):1319-1326. doi: 10.1007/s11606-020-06529-z. Epub 2021 Mar 10. PMID 33694071
- See also: Impact of the Early Phase of the COVID-19 Pandemic on US Healthcare Workers: Results from the HERO Registry — https://pubmed.ncbi.nlm.nih.gov/33694071/
- See also: Racial/Ethnic Disparities in Healthcare Worker Experiences During the COVID-19 Pandemic: An Analysis of the HERO Registry — https://pubmed.ncbi.nlm.nih.gov/35265822/
- See also: Patterns of Potential Moral Injury in Post-9/11 Combat Veterans and COVID-19 Healthcare Workers — https://pubmed.ncbi.nlm.nih.gov/35381899/
- See also: Gender and intention to leave healthcare during the COVID-19 pandemic among U.S. healthcare workers: A cross sectional analysis of the HERO registry — https://pubmed.ncbi.nlm.nih.gov/37327216/
- See also: Experiences of U.S. Nurses Compared With Nonnurses in the First Year of COVID-19: Findings From a National Registry — https://pubmed.ncbi.nlm.nih.gov/35878076/